## **Cover Page**

## **Statistical Analysis Plan**

Study Title: Equity Using Interventions for Pain and Depression (EQUIPD) - Phase 1

NCT05695209

**Document Date:** 1/27/2025

## **Data Analysis (Statistical Analysis Plan)**

Statistical Methods. Proportions were calculated for the number of participants who were retained at 3 and 6 months, as well as for those who completed at least 3 of the 4 coaching sessions (i.e., intervention adherence). Summary statistics were calculated overall and by treatment group for all demographic characteristics. Demographic characteristics were compared between treatment groups with appropriate statistical tests (i.e., Fisher's exact or Wilcoxon rank sum test) to verify that the randomization process produced balanced groups. Study outcomes were summarized by treatment group at each timepoint. Effect sizes were estimated using Hedge's g, which was calculated as follows: (change from baseline for intervention group - change from baseline for control)/mean standard deviation of change for each group at each timepoint. Hedge's g values of .20, .50, and .80 are typically interpreted as small, medium, and large effects, respectively. Analyses were conducted in SAS/STAT ® Software version 9.4 (SAS Institute Inc., Cary, North Carolina, USA).

## Reference

1. Hedges LV. Distribution theory for Glass's estimator of effect size and related estimators. *Journal of Educational Statustics*. 1981;6(2):107-28. doi:10.2307/1164588